CLINICAL TRIAL: NCT06429566
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase IIa Clinical Trial to Evaluate the Efficacy and Safety of Oral Local Use of GB001 Recombinant Peptide Spray for the Treatment of Mild Recurrent Aphthous Ulcer
Brief Title: Safety and Efficacy Study of GB001 Recombinant Peptide Spray in Subjects With Mild Recurrent Aphthous Ulcers
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Echon Biopharm Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YK2019L01P-IIa
Record Dates: First submitted 2024-04-30; First posted 2024-05-28 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GB001 recombinant peptide spray low dose group (Experimental): Each subject will take oral GB001 recombinant peptide spray 4 times a day, 4 sprays each time, no more than 29 times，The dosage of the group is 0.108mg/spray.
  Interventions: Drug: GB001 recombinant peptide spray low dose group、high dose group
- GB001 recombinant peptide spray high dose group (Experimental): Each subject will take oral GB001 recombinant peptide spray 4 times a day, 4 sprays each time, no more than 29 times，The dosage of the group is 0.216mg/spray.
  Interventions: Drug: GB001 recombinant peptide spray low dose group、high dose group
- Placebo group (Experimental): Each subject will take oral GB001 recombinant peptide spray 4 times a day, 4 sprays each time, for 8 days.
  Interventions: Drug: GB001 recombinant peptide spray placebo

INTERVENTIONS:
Drug: GB001 recombinant peptide spray low dose group、high dose group — Administrated oral spray. Each subject will take oral GB001 recombinant peptide spray 4 times a day, 4 sprays each time, no more than 29 times，The dosage of the group is 0.108mg/spray for low dose group and 0.216mg/spray for high dose group.
  Arms: GB001 recombinant peptide spray high dose group; GB001 recombinant peptide spray low dose group
Drug: GB001 recombinant peptide spray placebo — Administrated oral spray.Each subject will take oral GB001 recombinant peptide spray placebo 4 times a day, 4 sprays each time, no more than 29 times
  Arms: Placebo group

SUMMARY:
This trial is conducted in China. The purpose is to evaluate the efficacy, Pharmacokinetics (PK) profile, immunogenicity and safety of GB001 recombinant peptide spray in adults with mild recurrent aphthous ulcer.

ELIGIBILITY:
Inclusion Criteria:

1. It meets the diagnostic criteria for mild recurrent Aphthous ulcer in the fifth edition of Oral Mucosa published by People's Medical Publishing House in 2020.
2. 18≤ age ≤65 years old, gender is not limited.
3. Patients with untreated target ulcer onset ≤48 hours at the time of screening.
4. VAS score of target ulcer irritation pain ≥3 points, 2mm≤ length diameter of target ulcer ≤10mm.
5. Subjects and their sexual partners agree to use effective contraception during the study period and for at least 30 days after the study ends.
6. Sign a written informed consent, and be able to comply with the visit and related procedures stipulated in the program.

Exclusion criteria:

1. The diagnosis was severe aphthous ulcer, herpetic aphthous ulcer, acute herpetic gingivitis stomatitis, traumatic ulcer, cancerous ulcer, tuberculous ulcer, syphilitic ulcer, necrotic salivate metaplasia, Behcet disease and other diseases or drug induced ulcers.
2. Patients with suppurative tonsillitis or other painful lesions in the mouth, such as pericoronitis, pulpitis, periapical inflammation, etc., affecting the pain score of target ulcer.
3. Target ulcer is affected by residual root, residual crown, denture, prosthesis, orthodontic device and other stimulating factors in the corresponding parts of the target ulcer.
4. The ulcer is located in the lingual frenulum, the back wall of the pharynx and other parts, and its size is not easy to measure.
5. Those who plan to perform other oral treatments during the trial that affect the determination of drug effectiveness and safety.
6. Smokers > 20 cigarettes/day or betel nut lovers in the past 3 months.
7. People who have used painkillers or drugs that may affect the efficacy of pain observation within 24 hours before the first administration, such as sedatives, anti-allergy drugs, non-steroidal anti-inflammatory drugs, etc.
8. Patients who have used antibiotics or antiviral drugs locally or systematically within 1 week before screening.
9. Patients who had used immunosuppressive agents locally within 1 week before screening or systemic immunosuppressive agents within 2 weeks before screening.
10. Patients with oral local or systemic use of glucocorticosteroids within 4 weeks prior to screening.
11. Patients who have taken anticholinergic drugs to reduce salivary secretion within 2 weeks prior to screening.
12. Complicated with severe liver and kidney diseases, or abnormal liver and kidney function tests (ALT and AST≥ 1.5 times the upper limit of normal, SCr > the upper limit of normal).
13. Patients with severe anemia (Hb < 60g/L).
14. Complicated with severe heart and lung disease, uncontrolled diabetes (fasting blood glucose > 7.0mmol/L or random blood glucose ≥11.1mmol/L), advanced tumors, diseases of the blood and hematopoietic system, or other serious or progressive diseases of the system.
15. Known or suspected allergic history or serious adverse reactions to the experimental drug and its excipients.
16. Pregnant or lactating women and those with recent pregnancy plans.
17. Participants who had participated in other interventional clinical trials within 3 months prior to screening.
18. Other conditions deemed inappropriate by the investigator for participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-07-18 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
Target ulcer healing rate for patients in day 6 | Day 6
  Ulcer healing was defined as disappearance of pain and zeroing of ulcer size. At the screening visit the ulcer area and pain severity of patient to clinical examination will be rated at baseline. The patients will be self-assessment pain severity in vas score sheet every day . And the patients will be re-examined in day 6 to assess the ulcer area by periodontal probe.
Subjects self-rated the time it took for irritation pain to disappear | Day 8

SECONDARY OUTCOMES:
Time for target ulcer to heal | Day 8
  Ulcer healing was defined as disappearance of pain and zeroing of ulcer size.The patients will be self-assessment pain severity in vas score sheet every day . And the patients will be re-examined to assess the ulcer area by periodontal probe.
Targeted ulcer healing rate for patients in day 4 and day 8 | Day 4,Day 8
  Ulcer healing was defined as disappearance of pain and zeroing of ulcer size. At the screening visit the ulcer area and pain severity of patient to clinical examination will be rated at baseline. The patients will be self-assessment pain severity in vas score sheet every day . And the patients will be re-examined in day 4 and day 8 to assess the ulcer area by periodontal probe.
Changes in target ulcer area relative to baseline | Day 4,Day 6,Day 8
  At the screening visit the ulcer area of patient to clinical examination will be rated at baseline. And the patients will be re-examined in day 4、day 6 and day 8 to assess the ulcer area by periodontal probe.
Self evaluation of pain disappearance rate and relief rate | Day 4,Day 6,Day 8
Pharmacokinetics Characteristics， t½ of GB001 Recombinant Peptide | Day 1,Day 4
  Apparent terminal phase half-life
Pharmacokinetics Characteristics，AUC of GB001 Recombinant Peptide | Day 1,Day 4
  Area under the plasma concentration versus time curve
Pharmacokinetics Characteristics， Cmax of GB001 Recombinant Peptide | Day 1,Day 4
  Maximum plasma concentration
Pharmacokinetics Characteristics， Tmax of GB001 Recombinant Peptide | Day 1,Day 4
  Time of maximum plasma concentration
Immunogenicity(drug resistant antibody (ADA)) | Day 1,Day 14,Day 28
Incidence of Adverse Events | First dose to last visit,an average of 1 month.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Hunan University of Chinese Medicine, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No